CLINICAL TRIAL: NCT06518460
Title: Development and Testing of a New Tool for Evaluating Functional Self-sufficiency in Post-acute Stroke Patients
Brief Title: Functional Efficiency of Self-sufficiency Test
Acronym: FEST
Status: Completed | Type: Observational
Sponsor: Palacky University (Other)
Responsible Party: Principal Investigator, Jana Vyskotova, PhD., MSc., Palacky University
Other Study IDs: 61989592
Record Dates: First submitted 2024-03-24; First posted 2024-07-24 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Stroke/Brain Attack
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Functional Efficiency of Self-sufficiency Test — The Barthel Index has 10 items focusing on mobility, feeding, grooming, hygiene, dressing, bladder control and bowel control. It scores from 0-100 points. A higher score indicates better performance. The Action Research Arm Test is 19-item observational measure used for the assessment of UE performance in stroke recovery. Scores range from 0-57 points. A higher score indicates a better outcome.
  Other Names: The Barthel Index, The Action Research Arm Test

SUMMARY:
The aim of this study is to design and validate new tool for evaluation of self-sufficiency in post-acute stroke patients. And further identify the factors influencing changes in the Functional Efficiency of Self-sufficiency Test (FEST) in post-acute rehabilitation care.

DETAILED DESCRIPTION:
The research included the development of the FEST and its validation and the determination of the influence of selected factors on the change in functional self-sufficiency assessed by FEST.

The FEST consists of nine assessed categories (mobility, stability, locomotion, dressing, hygiene, eating, household care, communication, finances), which allow a comprehensive assessment of the current status of post-acute stroke patients. Patients meeting inclusion criteria are screened: 1/ diagnosed with ischemic or haemorrhagic stroke in the post-acute stage; 2/ aged ≥18 years; 3/ stable vital functions; 4/ rehabilitation load of 4 hours per day; 5/ maintained swallowing functions. Exclusion criteria: 1/ tracheostomy; 2/ not recommended by psychotherapist due to cognitive deficit and unwillingness; 3/ severe sensory deficit (hearing, vision). Patients are tested at the beginning (first measurement) and at the end of the post-acute rehabilitation care (second measurement) at the rehabilitation institute. The battery of tests included FEST, BI, the Action Research Arm Test (ARAT).

Descriptive statistics will use for the basic statistical analysis. Cronbach's alpha will use to assess reliability. The correlation between variables will calculate using Spearman's and Pearson's correlation coefficients and the biserial correlation coefficient. Construct validity will assess using factor analysis. The difference between independent samples will verify by two-sample t-test. The effect of baseline demographic characteristics (age, gender), and UA functional status on the improvement in the level of self-sufficiency measured by FEST will verify by multivariate linear regression. All tests will perform at a significance level of 0.05. IBM SPSS Statistics for Windows (version 23.0) statistical software will use for statistical processing (Armonk, NY: IBM Corp).

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with ischemic or haemorrhagic stroke in the post-acute stage; aged ≥18 years; stable vital functions; rehabilitation load of 4 hours per day; maintained swallowing functions.

Exclusion Criteria:

* tracheostomy; not recommended by psychotherapist due to cognitive deficit and unwillingness; severe sensory deficit (hearing, vision).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: post-acute stroke adult patients
Sampling Method: Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Psychometric characteristics validation | 1.8.2024-31.8.2025
  The following tests will be performed on the FEST test: internal consistency, correlation between variables, convergent validity, and factor analysis. The psychometric properties of the FEST will be compared with those of the Barthel Index and the Action Research Arm Test.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Kisvetrova, Study Director — Palacky University Olomouc
Locations (1):
- Palacky University, Olomouc, Czech, Czechia

IPD SHARING:
Plan to Share IPD: No